CLINICAL TRIAL: NCT02307799
Title: A RESearch on the PrEvalence and the Diagnosis of COPD and Its Tobacco-related Etiology (RESPECT)
Brief Title: A RESearch on the PrEvalence and the Diagnosis of COPD and Its Tobacco-related Etiology
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Jean-Marie Degryse, professor, Université Catholique de Louvain
Other Study IDs: RESPECT2014
Record Dates: First submitted 2014-11-26; First posted 2014-12-04 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: tobacco; spirometry; cohort study; case-control study; prevalence
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the RESPECT study is to gain a better understanding of the prevalence, pathogenesis and symptoms of early chronic obstructive pulmonary disease (COPD). This study seeks to address the following specific objectives/research questions: 1) to estimate the prevalence of airflow limitation (AL) and COPD in adults 35-70 years of age in St.Petersburg and Arkhangelsk based on sex, age, environmental conditions, socioeconomic status and smoking status; 2) to compare the prevalence of COPD in the study population based on the Global Strategy for Diagnosis, Management and Prevention of COPD (GOLD) and lower limit of normal (LLN) criteria; 3) to identify the diagnostic value of various signs, symptoms and background characteristics for the diagnosis of COPD; 4) to determine whether differences in background characteristics and inflammatory biomarkers are evident between smokers with and without COPD; and 5) to describe co-morbidity, functionality and global health status in a cohort of newly diagnosed COPD patients.

DETAILED DESCRIPTION:
Two northwestern of Russian Federation (RF) cities (St.Petersburg and Arkhangelsk) were selected for the RESPECT study. Fifteen primary care centers were invited to participate in this study.

Fifteen investigators (10 from St.Petersburg and 5 from Arkhangelsk) were recruited (predominantly doctors and two highly educated nurses). All investigators received study information, including a detailed study protocol and recent guidelines on COPD, and participated in a three-week course on spirometry and the clinical diagnosis and management of obstructive lung diseases. The sample size was calculated based on two goals: 1) to determine a reliable estimate of the prevalence of COPD and 2) to estimate the diagnostic value of symptoms with an acceptable confidence interval.

The sample size for the RESPECT study was estimated using 2828 subjects (based on an 8% prevalence of COPD in RF). Assuming an anticipated refusal rate of 20%, 3500 participants from St.Petersburg and 1500 from Arkhangelsk were invited to participate in this study.

The analyses will include cross-sectional and prospective approaches. Prospective analyses will be performed on the entire cohort.

ELIGIBILITY:
Inclusion Criteria:

•written consent to participate

Inclusion criteria for the cohort component:

•100 newly detected persons with FEV1/FVC less than 0.7 or less than LLN before and after reversibility test.

Inclusion criteria for the case-control component:

Both for cases and controls:

•A smoking history of more than 10 pack-years based on pack/year criteria

Test cases will include 100 participants that meet the following criteria:

* Smokers aged 35-70 years with a smoking history of >10 pack-years.
* Completely irreversible airway obstruction based on the following criteria: FEV1/FVC < 0.70 according to GOLD criteria or FEV1/FVC < LLN.

Test controls will include 100 participants based on the following criteria:

•Smokers aged 35-70 years with a smoking history of >10 pack/years and without COPD according to GOLD or LLN criteria, without asthma (absence of symptoms), with a negative history of allergies, and free from use of bronchodilators.

Exclusion Criteria:

* COPD exacerbation during last 3 months
* Patient did not sign an informed consent
* Patient refuses to participate

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First component: The study population was randomly selected from the lists of the 15 participating centers (these patient lists are organized based on territories).
  Second component (cohort study): All newly identified individuals with airflow limitation before and/or after the reversibility test were included in the cohort study.
  Third component: One hundred patients with COPD and a smoking history of more than 10 pack-years (cases) and one hundred patients with the same smoking history without COPD (controls) will be included in the third study.
Sampling Method: Probability Sample
Enrollment: 3133 (Actual)
Dates: Start 2012-06; Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change of lung function parameter (FEV1/FVC (Forced Vital Capacity) and FEV1) | Change from Baseline FEV1/FVC and FEV1 at 1 year
  Evolution of lung function parameters

SECONDARY OUTCOMES:
Change of positive predictive value of signs and symptoms | Change from Baseline signs and symptoms at 1 year
  diagnostic value of signs and symptoms (positive predictive value)
Change of inflammatory parameters | Change from Baseline inflammatory parameters at 1 year
  inflammatory profiles (biomarkers)
Comorbidities (comorbidities for COPD) | Change from Baseline number of comorbidities at 1 year
  number of comorbidities for COPD
Change of health status (The change in health status by the Questionnaire of the EuroQol Group Association) | Change from Baseline Health Status at 1 year
  The change in health status by the Questionnaire of the EuroQol Group Association

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Degryse, professor, Principal Investigator — Université Catholique de Louvain, Brussels, Belgium; Olga Yu Kuznetsova, professor, Principal Investigator — North-West State Medical University, St Petersburg, Russia; Elena A Andreeva, PhD, Principal Investigator — Northern State Medical University, Arkhangelsk, Russia; Marina A Pokhaznikova, PhD, Principal Investigator — North-West State Medical University, St Petersburg, Russia
Locations (2):
- Russia (2):
  - City Policlinic Number 2, Arkhangelsk
  - Family medicine center, Saint Petersburg

REFERENCES:
- [Background] Andreeva E, Pokhaznikova M, Lebedev A, Moiseeva I, Kozlov A, Kuznetsova O, Degryse JM. The RESPECT study: RESearch on the PrEvalence and the diagnosis of COPD and its Tobacco-related etiology: a study protocol. BMC Public Health. 2015 Aug 28;15:831. doi: 10.1186/s12889-015-2161-z. PMID 26315949
- [Result] Andreeva E, Pokhaznikova M, Lebedev A, Moiseeva I, Kutznetsova O, Degryse JM. The Prevalence of Chronic Obstructive Pulmonary Disease by the Global Lung Initiative Equations in North-Western Russia. Respiration. 2016;91(1):43-55. doi: 10.1159/000442887. Epub 2016 Jan 5. PMID 26727503
- [Result] Andreeva E, Pokhaznikova M, Lebedev A, Moiseeva I, Kuznetsova O, Degryse JM. Spirometry is not enough to diagnose COPD in epidemiological studies: a follow-up study. NPJ Prim Care Respir Med. 2017 Nov 14;27(1):62. doi: 10.1038/s41533-017-0062-6. PMID 29138407
- [Derived] Andreeva E, Pokhasnikova M, Lebedev A, Moiseeva I, Kozlov A, Kuznetsova O, Degryse JM. Inflammatory parameters and pulmonary biomarkers in smokers with and without chronic obstructive pulmonary disease (COPD). J Thorac Dis. 2021 Aug;13(8):4812-4829. doi: 10.21037/jtd-20-1580. PMID 34527321